CLINICAL TRIAL: NCT05335239
Title: Domiciliary Professional Cleaning for Care Dependent Older Adults - A Randomized Controlled Trial
Brief Title: Domiciliary Professional Oral Care for Dependent Older Adults
Acronym: HET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Inger Wårdh, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KarolinskaDalarnaGävleborg
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2023-06

CONDITIONS: Dental Caries of Root Surface; Aging
Keywords: Dental prophylaxis; Aged; Dental devices, Home Care; Root Caries; Sodium Fluoride
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Single - blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Every third month, a dental assistant will visit at home and deliver professional dental cleaning and delivery of one new toothbrush and fluoride toothpaste (>4000ppm) (n:3) for the next three months. The visit is expected to take at the most 30 minutes.
  Interventions: Other: Professional dental cleaning
- Controll group (No Intervention): Continuous with oral care as usual, either by themselves or nursing assisted (help with oral hygiene procedure) during the whole study period. Home care aides working with the control study participants delivers a toothbrush and fluoride toothpaste (> 4000 ppm) (n:3) every third month during the study period.

INTERVENTIONS:
Other: Professional dental cleaning — The dental assistant will visit at home and delivers professional dental cleaning, a reminder to use the fluoridated toothpaste (> 4000 ppm ) and oral hygiene instruction to participants accompanied by home care aides, with manual toothbrush, fluoridated toothpaste (> 4000 ppm) and relevant interproximal aids.
  Arms: Intervention group

SUMMARY:
Keep brushing your teeth, twice a day, during life for healthy teeth and body. Not brushing your teeth regularly and well, may have a devastating effect on your teeth and your general health. The teeth could develop root caries resulting in pain, fractured teeth, tooth loss and trouble eating. Further, brushing your teeth insufficiently leads to higher number of bacteria in the oral cavity and could in frail individuals lead to aspirations pneumonias.

With age, some of us will depend on daily care activities from others and help with daily toothbrushing. However, care dependent older adults often lack basic dental care (tooth brushing with fluoride tooth paste twice a day).

Dental care at home is a service proved by dental personnel. Visits at a dental clinic decrease with age and especially with a dementia diagnosis. Dental care at home can deliver regular dental check-ups and dental treatments to individuals who experience difficulties attending a dental clinic.

The effect of teeth cleaning performed at home on root caries development, has not yet been explored in care dependent older adults. Therefore, the aim is to study if the combination of high fluoride toothpaste used daily with teeth cleaning/ a reminder to use the toothpaste every third month, could be a method for preventing root caries development in this patient group.

The hypothesis is that domiciliary professional cleaning will improve the oral health, as measured by root caries development, gingival bleeding, plaque accumulation and oral mucosal status, compared with a control group that receives oral care as usual.

DETAILED DESCRIPTION:
Care dependent older adults living in nursing homes have high rates of untreated root caries lesions (RCLs). RCLs, if left untreated could lead to pain, tooth loss, difficulties eating, and impacts on general health. An increasing number of research publications point to the association between poor oral health, respiratory tract infections and aspiration pneumonia. Therefore, there is a need for prevention and effective treatment among older adults, and especially those who are care dependent.

When hospitalized or being care dependent, help with care often depends on others. However, nursing assisted oral care/help with oral hygiene, is a difficult task. An effective method for preventing and treating RCLs is to brush the teeth twice a day with high fluoride toothpaste containing 5000 ppm F - . Toothpaste containing 5,000 ppm F - decreases the numbers of RCLs in comparison with ordinary toothpaste containing 1,100 - 1,450 ppm F - .

Visits at a dental clinic decrease with age and especially with a dementia diagnosis. For that reason, the service domiciliary dental care (DDC), could be an option since DDC enables dental care at home (check-ups, prophylaxis, simple tooth extractions, tooth restorations and prothesis adjustments) by dental personnel. DDC could be beneficial for the older adults, due to not having to leave home.

The effect of DDC on root caries development, has not yet been explored in care dependent older adults.

Objectives: The aim is to evaluate the effects of domiciliary professional cleaning for care dependent home living older adults. Furthermore, to contribute to increased knowledge for establishing oral health care recommendations about frequency and content for domiciliary preventive professional oral care in this patient group.

The first hypothesis is that domiciliary professional cleaning will improve the oral health, as measured by; root caries development, gingival bleeding, plaque accumulation and oral mucosal status, compared with a control group that receives assisted oral care as usual.

The second hypothesis is that domiciliary professional cleaning will improve the general health status, as measured by; oral health related quality of life, number of antibiotic treatments and number of respiratory tract infections, compared with a control group that receives assisted oral care as usual.

Study design: The project is designed as a randomized control trial (RCT), evaluator blinded, with two parallel study arms for one year. Randomization will be performed at individual level by a person not otherwise involved in the project.

Data collection will be performed at baseline and at twelve months, by calibrated registered dental hygienists (RDH) assisted by dental assistants. For the intervention, two additional dental assistants, will visit the study participants. Data analysis will be presented at group level and dropouts will be handle according to per protocol analysis.

Description of the study population: Variables regarding cognitive functions by Pfeiffer's test, age, gender, number of respiratory tract infections, oral hygiene habits (frequency of toothbrushing, performing oral hygiene routine by themself or nursing assisted oral care, frequency of interproximal cleaning), dental status (number of teeth, root tips, fillings, dental caries, missing teeth, implants) and drug intake (gathered from responsible nurse) will be collected during baseline visit for descriptive measurements.

The sample size is based on a power calculation (two-tailed) for the primary effect variable root caries, 63 individuals in each group are required. Due to high drop-out rates previously reported in the study population, the sample will be increased by 25%. Accordingly, the number of participants will be n=158 (79 in each group).

Data registration:

* Dental root caries lesions
* Gingival bleeding/Bleeding on probing (BoP)
* Oral hygiene
* Oral health related quality of life
* General health
* Oral microbiota: Collection of dental plaque and unstimulated saliva samples will be performed single-blinded in a subsample of 50 from the total study population. To possibly elucidate the causes behind the oral health situation. The PhD-student is responsible for coding, adequate storage and the transport to the lab for analysis. Analysis of saliva samples will be performed at NGS at the appropriate core facilities (SciLifeLabs) at Karolinska Institutet (Professor Belibasakis). Dental plaque at Umeå University, Institute of Odontology, Clinical Oral Microbiology Laboratory (Dr. Anders Johansson). All samples will, after completion of the process at the lab (up to six months after collection), be destroyed.

The participants are consecutively recruited during their annually oral health assessments and sorted to intervention or control group after informed consent. All study participants will, after baseline, start with fluoridated toothpaste ≥ 4000 part per million (ppm) for brushing their teeth twice a day during the study period to establish an equivalent oral hygiene routine. For controlling the adherence to the toothpaste routine, all participants will receive a litterbox to throw empty toothpaste tubes during the study period.

Preliminary results: The previous study was a RCT - study performed at nursing homes during six months. The intervention group received monthly professional dental cleaning, oral hygiene information and instruction, by RDHs. The control group continued with oral care as usual. Data collection was performed every third month. The analysis showed an improvement in both groups for gingival bleeding, mucosal score and root caries. Due to improvement in both groups, the upcoming study will reduce the prophylactic visits to every third month. Reducing visits is economical beneficial since delivering home care is often more time consuming. Also, instead of having RDHs for the visits, we now engage dental assistants. Dental assistants have prophylactic training in their education and it is important that every profession have possibilities to fully take advantage of their competence.

Significance: Oral diseases and especially dental root caries are common among older adults and increase with age. Among care dependent older adults the amount of untreated root caries is high, causing (if left untreated) pain, tooth loss and impacts on general health. An increasing number of research publications point to the association between poor oral health, aspiration pneumonia and quality of life. For that reason, the need for prevention and effective treatments for root caries is important among older adults, and especially those who need help with daily activities. For prevention, one simple and effective method is to use fluoride toothpaste containing 5000 ppm NaF daily. The combination with this toothpaste and prophylactic/reminding home visits every third month by a dental assistants, could be an effective method for preventing root caries in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Home-living older adults
* Age ≥65
* Eligible for subsidized dental care for those with in-home care
* Accepted oral health assessment by dental hygienists
* Non-smokers
* Ability to cooperate during oral assessment for 5-10 minutes
* At least one natural tooth
* Understand and able to communicate in Swedish.
* Additionally: For oral microbiota, grade 1-2 according to mirror slide friction test.

Exclusion Criteria:

* Edentulousness
* Full dentures
* Cognitive limitations that is an obstacle for cooperation
* Malignancies and/or immunosuppressive diseases
* Coagulation defects.
* Anticoagulants are registered but not as an exclusion criterion.
* Moving or planned to move to a nursing home
* For oral microbiota: grade 3 according to mirror slide friction test

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Dental root caries | 12 months
  Registered by the Fejerskov´s five levels root caries index at baseline and after twelve months.

SECONDARY OUTCOMES:
Oral health-related quality of life | 12 months
  Measured by Geriatric Oral health Assessment GOHAI at baseline and after twelve months.
Oral hygiene | 12 months
  Measured by mucosal and plaque index, MPS and will be used both for fixed teeth and removable prosthesis, at baseline and twelve months.
Gingival bleeding | 12 months
  Bleeding on probing (BoP) in the gingival sulcus on buccal surfaces using the Ramfjord teeth (RT) 16, 21, 24, 36, 41, 44 or the nearest comparable teeth. The bleeding will be scored at four levels (0-3) due to Modified Sulcus Bleeding Index at baseline and after twelve months.
Oral microbiota | 12 months
  To possibly elucidate the causes behind the oral health situation. Collection of dental plaque and unstimulated saliva samples will be performed single-blinded in a subsample of 50 in the study population at baseline and after twelve months.
General health | 12 months
  Number of episodes with respiratory tract infections, pneumonia and use of antibiotics. Data is collected from medical responsible nurses at baseline and after twelve months.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Wårdh, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska institute, Huddinge, Sweden

REFERENCES:
- [Result] Girestam Croonquist C, Dalum J, Skott P, Sjogren P, Wardh I, Moren E. Effects of Domiciliary Professional Oral Care for Care-Dependent Elderly in Nursing Homes - Oral Hygiene, Gingival Bleeding, Root Caries and Nursing Staff's Oral Health Knowledge and Attitudes. Clin Interv Aging. 2020 Aug 6;15:1305-1315. doi: 10.2147/CIA.S236460. eCollection 2020. PMID 32982191
- See also: Fulltext Girestam et al 2020 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7495352/pdf/cia-15-1305.pdf